CLINICAL TRIAL: NCT03050554
Title: Phase I/II Study of the Safety, Tolerability, and Efficacy of Stereotactic Body Radiation Therapy (SBRT) Combined With Concurrent and Adjuvant Avelumab for Definitive Management of Early Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: SBRT Combined With Avelumab (Anti-PD-L1) for Management of Early Stage Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Andrew Sharabi (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Andrew Sharabi, Assistant Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161591
Record Dates: First submitted 2017-02-02; First posted 2017-02-13 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Early Stage Non-Small Cell Lung Cancer
Keywords: cancer; Non-Small Cell Lung Cancer; SBRT; Avelumab; Stereotactic Body Radiation Therapy; radiation; NSCLC; PD-1; PD-L1; Immunotherapy; Lung
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SBRT+Avelumab (Experimental): SBRT: 12Gy x 4 fractions or 10Gy x 5 fractions (4-5 radiation doses given over 10-12 days every other day.)
  Avelumab 10mg/kg IV infusion every 2 weeks for 6 cycles
  Interventions: Drug: Avelumab; Radiation: SBRT

INTERVENTIONS:
Drug: Avelumab — Avelumab 10mg/kg IV infusion every 2 weeks for 6 cycles
  Other Names: Bavencio
Radiation: SBRT — SBRT: 12Gy x 4 fractions or 10Gy x 5 fractions (4-5 radiation doses given over 10-12 days every other day.)
  Other Names: Stereotactic Body Radiation Therapy

SUMMARY:
The purpose of the study is to determine whether avelumab has an effect on cancer and body in combination with SBRT, a standard treatment for early stage non-small cell lung cancer (NSCLC).

Avelumab is considered experimental because it is not approved by the United States (U.S.) Food and Drug Administration (FDA) for the treatment of cancer. It is a type of drug called a monoclonal antibody (a type of protein). Monoclonal antibodies are made to recognize, target and bind to specific proteins on the cells that make up your tissues. Avelumab is designed to block the interaction between PD-1, a known immune checkpoint, and PD-L1. By blocking this interaction, the immune system may be stimulated, allowing it to more effectively recognize and attack the cancer.

Stereotactic Body Radiation Therapy (SBRT) is a type of radiation that uses precise targeting to deliver a high dose of radiation to the tumor over a short period of time. A positioning cushion such as Vac-lok will be used during radiation treatment that is custom made. This custom mold forms to the contours of the subjects body to allow for proper positioning comfort and stability.

DETAILED DESCRIPTION:
This is a single arm open label Phase I/II study that will consist of two parts. In Phase I, investigators will assess the safety and tolerability of SBRT combined with Avelumab. In Phase II, investigators will determine whether SBRT combined with Avelumab improves relapse free survival. Subjects with Stage I NSCLC who are not undergoing surgical resection will be candidates for enrollment. Subjects will receive definitive stereotactic body radiation (SBRT) in 4-5 fractions combined with concurrent and adjuvant Avelumab at 10mg/kg for a total of 6 cycles. Subjects will be evaluated for safety as measured by the occurrence of adverse events, serious adverse events, and laboratory abnormalities. Three blood draws will be obtained to analyze anti-tumor immune responses and immune correlates.

ELIGIBILITY:
Inclusion Criteria:

* Tumor(s) to be treated is(are) ≤ 5.0 cm or ≤250 cm3
* Stage I NSCLC and is deemed medically inoperable or refuses surgical resection.
* Life expectancy ≥ 9 months.
* Acceptable organ and marrow function

Exclusion Criteria:

* Prior organ transplantation, including allogeneic stem cell transplantation
* Significant acute or chronic infections including:

  * Known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
  * Known history of HBV or HCV
* Active autoimmune disease

  * Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
  * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
  * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
* Current use of immunosuppressive medication, EXCEPT for the following:

  * intranasal, inhaled, topical steroids, or local steroid injection (eg, intra-articular injection)
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure, or serious cardiac arrhythmia requiring medication.
* Known severe hypersensitivity reactions to monoclonal antibodies any history of anaphylaxis, or uncontrolled asthma
* Pregnancy or lactation
* Known alcohol or drug abuse
* Prior radiotherapy to the treatment site(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sharabi, M.D., Ph.D., Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Sanford Health, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT+Avelumab: SBRT: 12Gy x 4 fractions or 10Gy x 5 fractions (4-5 radiation doses given over 10-12 days every other day.)
  Avelumab 10mg/kg IV infusion every 2 weeks for 6 cycles
  Avelumab: Avelumab 10mg/kg IV infusion every 2 weeks for 6 cycles
  SBRT: SBRT: 12Gy x 4 fractions or 10Gy x 5 fractions (4-5 radiation doses given over 10-12 days every other day.)
Period: Overall Study
Arm/Group | SBRT+Avelumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SBRT+Avelumab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Safety and tolerability of definitive SBRT combined with concurrent and adjuvant Avelumab in patients with early stage NSCLC (Measured Via Adverse Events).
Time Frame: 6 months
Population: The study was terminated due to low enrollment and difficulty with accrual. We accrued 2 patients in 1 year and then Pfizer who was supported the study pulled their funding. So then the study was unfunded and needed to be terminated.
Arm/Group | SBRT+Avelumab
Number analyzed (Participants) | 0

2. Primary Outcome: Relapse Free Survival (RFS)
Description: Relapse-Free Survival (RFS) is defined as the time from starting treatment to the time of first documented tumor progression or death due to any cause, whichever occurs first. Death is considered as an event here.
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | SBRT+Avelumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Loco-regional Control (LRC)
Description: Locoregional Control (LRC) is defined as the time from starting treatment until local and/or regional relapse is documented
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | SBRT+Avelumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival in Patients After Completion of SBRT in Combination With Avelumab
Description: Overall survival in patients is defined as the time from after completion of SBRT in combination with Avelumab
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | SBRT+Avelumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | SBRT+Avelumab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT+Avelumab (N=2)
Cholecystitis (Gastrointestinal disorders) | 1 (1) — Cholecystitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT+Avelumab (N=2)
Fatigue (General disorders) | 2 (6) — Fatigue
Left Rib Pain with Deep Inspiration (Musculoskeletal and connective tissue disorders) | 1 (1) — Left Rib Pain with Deep Inspiration
Infusion Reaction (General disorders) | 1 (5) — Infusion reaction
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Cough
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Right Eye Pain and Redness (Eye disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1) — Right eye
Paresthesia (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Black Skin Tags (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03050554/Prot_SAP_002.pdf